CLINICAL TRIAL: NCT07270393
Title: Estudio de la Influencia de la Dieta mediterránea en la Calidad de Vida de Las Pacientes Con Endometriosis.
Brief Title: Study of the Influence of the Mediterranean Diet on the Quality of Life of Patients With Endometriosis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PAR-DON-2024-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis
Keywords: Endometriosis; Mediterranean diet; Quality of life
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will not receive normocaloric Mediterranean diet recommendations.
- Intervention Group (Experimental): This group will receive a series of normocaloric Mediterranean diet recommendations.
  Interventions: Other: Diet supplementation

INTERVENTIONS:
Other: Diet supplementation — The severities of chronic disease symptoms correlate with the levels of analytical parameters of inflammation. Studies have been published in which the Mediterranean diet has an anti-inflammatory phenomenon, decreasing inflammation parameters. This decrease correlates with an improvement in symptoms .
  Endometriosis is a chronic inflammatory disease and the influence of the Mediterranean diet on the decrease of inflammation parameters in women with endometriosis has been studied.
  Arms: Intervention Group

SUMMARY:
The severities of chronic disease symptoms correlate with the levels of analytical parameters of inflammation. Studies have been published in which the Mediterranean diet has an anti-inflammatory phenomenon, decreasing inflammation parameters. This decrease correlates with an improvement in symptoms.

Endometriosis is a chronic inflammatory disease and the influence of the Mediterranean diet on the decrease of inflammation parameters in women with endometriosis has been studied.

The studies carried out to assess whether this decrease in inflammatory parameters correlates with clinical improvement and quality of life in these patients have low/very low scientific evidence (small sample size, no control group) and with different interventions (diets, restrictions and/or supplements), which prevent their analysis as a whole.

Therefore, our hypothesis is that the Mediterranean diet, due to its anti-inflammatory effect, can improve the symptomatology and quality of life of patients with endometriosis.

ELIGIBILITY:
INCLUSION CRITERIA:

* Female.
* Age 18-45.
* Premenopausal status.
* Radiological diagnosis (by transvaginal ultrasound and/or MRI) and/or surgical diagnosis of endometriosis.
* Follow-up in the Gynecology Department of OSI Donostia (at least 1 visit in the last year).
* Clinical score of at least 3/10 on the Numerical Scale in at least one symptom related to endometriosis).
* Possibility of understanding Spanish.
* Possibility of understanding the indicated dietary recommendations.
* Acceptance of inclusion in clinical study, by signing informed consent.

EXCLUSION CRITERIA:

* Diagnosis of Eating Disorder.
* Diagnosis of malabsorptive syndromes: Chron's disease, Ulcerative colitis, short bowel syndrome, gastric by-pass, irritable bowel.
* Other concomitant diseases that produce CPD.
* Autoimmune diseases.-
* Metabolic diseases requiring follow-up of specific diets.
* Diagnosed gluten intolerance.
* Vegan diet.
* Follow-up by a nutritionist.
* Diagnosis of severe mental illness requiring treatment.
* Pregnancy or current breastfeeding.
* Active cancer process.
* Personal history of gynecologic or digestive oncologic process.
* Change of treatment or surgery during follow-up.
* Surgery related to endometriosis or change of treatment in the 6 weeks prior to enrollment in the study.
* Drug abuse. Opioid analgesia < 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life and endometriosis. | 24 weeks
  Endometriosis Health Profile 30 (EHP-30) questionnaire (0-100)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Pain with menstruation or Dysmenorrhea - A numeric scale (0-10)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Pain with sexual intercourse or Dyspareunia - A numeric scale (0-10)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Pain with defecation or Dyschezia - A numeric scale (0-10)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Pain with urination or Dysuria - A numeric scale (0-10)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Non-menstrual pelvic pain - A numeric scale (0-10)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Abdominal bloating or distension - A numeric scale (0-10)
Pain intensity in symptoms related to endometriosis | 24 weeks
  Tiredness - A numeric scale (0-10)

SECONDARY OUTCOMES:
General Quality of Life | 24 weeks
  WHOQOL-BREF questionnaire. (0-100)
Use of analgesics | 24 weeks
  Collecting the use of analgesics.
Change in BMI | 24 weeks
  Abdominal and hip circumference. (cm)
Diet quality | 24 weeks
  Diet Quality Assessment Survey developed by the Spanish Society of Dietetics and Food Sciences (SEDCA).
Adherence to the Mediterranean diet | 24 weeks
  Diet adherence test, used in the PREDIMED study, available free of charge on the website of the Spanish Society of Dietetics and Food Sciences (SEDCA).
Satisfaction Survey | 24 weeks
  Brief questionnaire that seeks to know the patient's opinion about his or her experience and degree of satisfaction with different aspects of the study.

OTHER OUTCOMES:
Personal data | 24 weeks
  Date and place of birth.
Personal data | 24 weeks
  Number of children.
Physical examination | 24 weeks
  Weight (kg)
Physical examination | 24 weeks
  Height (cm)
Physical examination | 24 weeks
  Body Mass Index (BMI) (kg/m2)
Physical examination | 24 weeks
  Abdominal circumference. (cm)
Physical examination | 24 weeks
  Hip circumference (cm)
Obstetric history | 24 weeks
  Assisted reproduction treatments (Current/completed/future)
Obstetric history | 24 weeks
  Gestational desire
Medical history related to endometriosis | 24 weeks
  Type of endometriosis (Not reported/ Ovarian endometriosis/ Deep endometriosis/ Endometriosis)
Medical history related to endometriosis | 24 weeks
  Diagnosis of endometriosis by: radiology and/or surgery.
Medical history related to endometriosis | 24 weeks
  Previous diets performed.
Medical history related to endometriosis | 24 weeks
  Treatments received: Medical (hormonal contraception, analogues, other).
Medical history related to endometriosis | 24 weeks
  Treatments received: Surgical (conservative vs. radical surgery).
Current situation related to endometriosis | 24 weeks
  Symptoms.
Current situation related to endometriosis | 24 weeks
  Current treatment.
Medical history related to endometriosis | 24 weeks
  Diagnosis: Date- time of evolution since onset of symptom.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Donostia (HUD), Donostia / San Sebastian, Gipuzkoa, Spain